CLINICAL TRIAL: NCT03218566
Title: A Prospective, Multicenter Trial to Evaluate the Safety and Efficacy of the Indigo® Aspiration System in Acute Pulmonary Embolism
Brief Title: Evaluating the Safety and Efficacy of the Indigo® Aspiration System in Acute Pulmonary Embolism
Acronym: EXTRACT-PE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11373
Record Dates: First submitted 2017-07-06; First posted 2017-07-14 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; clot
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Other): Single Arm - Use of Indigo Aspiration System (mechanical thrombectomy) to treat pulmonary embolism
  Interventions: Device: Indigo Aspiration System

INTERVENTIONS:
Device: Indigo Aspiration System — use of mechanical thrombectomy to treat pulmonary embolism

SUMMARY:
To determine the safety and efficacy of the Indigo Aspiration System for aspiration mechanical thrombectomy in patients with acute pulmonary embolism (PE)

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs and symptoms consistent with acute PE with duration of 14 days or less. Evidence of PE must be from CTA.
* Systolic BP ≥ 90 mmHg with evidence of dilated RV with an RV/LV ratio > 0.9
* Patient is 18 years of age or older

Exclusion Criteria:

* tPA use within 14 days prior to baseline CTA
* Systolic BP < 90mmHg for 15min or the requirement of inotropic support to maintain systolic BP ≥ 90 mmHg
* Pulmonary hypertension with peak PA > 70 mmHg by right heart catheterization
* History of severe or chronic pulmonary hypertension
* Fi02 requirement > 40% or >6 LPM to keep oxygen saturations >90%
* Hematocrit < 28%
* Platelets < 100,000µL
* Serum creatinine > 1.8 mg/dL
* INR > 3
* aPTT (or PTT) > 50 seconds on no anticoagulation
* History of heparin-induced thrombocytopenia (HIT)
* Contraindication to systemic or therapeutic doses of anticoagulants
* Major trauma < 14 days
* Presence of intracardiac lead
* Cardiovascular or pulmonary surgery within last 7 days
* Cancer requiring active chemotherapy
* Known serious, uncontrolled sensitivity to radiographic agents
* Life expectancy < 90 days
* Female who is pregnant
* Intracardiac Thrombus
* Patients on ECMO
* Current participation in another investigational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akhilesh Sista, MD, Principal Investigator — NYU-Langone School of Medicine
Locations (22):
- United States (22):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - St. Joseph Health Hospital, Orange, California
  - Christiana Care, Newark, Delaware
  - Baptist Hospital of Miami, Miami, Florida
  - AdventHealth Tampa, Tampa, Florida
  - Grady Health System, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Our Lady of the Lake Hospital Inc., Baton Rouge, Louisiana
  - Detroit Medical Center, Detroit, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mercy Hospital South, St Louis, Missouri
  - New York University (NYU) Langone Medical Center, New York, New York
  - Mount Sinai, New York, New York
  - North Carolina Heart and Vascular Research (NCHVR), Raleigh, North Carolina
  - University of Pennsylvania Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Sanford Health, Sioux Falls, South Dakota
  - Sentara Vascular Specialists, Norfolk, Virginia
  - Charleston Area Medical Center (CAMC), Charleston, West Virginia

REFERENCES:
- [Derived] Jorge JV, Barreiros CA, Silva D, Cale R, Ribeiro JM. Extracorporeal mechanical support and aspiration thrombectomy in treatment of massive pulmonary embolism: a case report. Rev Bras Ter Intensiva. 2022 Oct-Dec;34(4):524-528. doi: 10.5935/0103-507X.20220342-pt. Epub 2023 Mar 3. PMID 36888834
- [Derived] Sista AK, Horowitz JM, Tapson VF, Rosenberg M, Elder MD, Schiro BJ, Dohad S, Amoroso NE, Dexter DJ, Loh CT, Leung DA, Bieneman BK, Perkowski PE, Chuang ML, Benenati JF; EXTRACT-PE Investigators. Indigo Aspiration System for Treatment of Pulmonary Embolism: Results of the EXTRACT-PE Trial. JACC Cardiovasc Interv. 2021 Feb 8;14(3):319-329. doi: 10.1016/j.jcin.2020.09.053. Epub 2021 Jan 13. PMID 33454291

RESULTS

PARTICIPANT FLOW:
Groups:
- Indigo Aspiration System: Single Arm - Use of Indigo Aspiration System (mechanical thrombectomy) to treat pulmonary embolism
  Indigo Aspiration System: use of mechanical thrombectomy to treat pulmonary embolism
Period: Overall Study
Arm/Group | Indigo Aspiration System
Started | 119
Completed | 110
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 73
  >=65 years | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.8 (14.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 103
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 37
  White | 72
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 119
BMI-Females [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI specific to female population.
  kg/m^2
    number analyzed (Participants) | 53
    (all) | 36.7 (10.39)
BMI-Males [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI specific to male population.
  kg/m^2
    number analyzed (Participants) | 66
    (all) | 31.7 (6.60)

OUTCOME MEASURES:

1. Primary Outcome: Right Ventricle/Left Ventricle (RV:LV) Ratio
Description: Change in RV/LV ratio per CTA
Time Frame: from baseline to 48 hours
Population: The intent-to-treat population calculating the change between the baseline and the 48 hours RV/LV diameter ratio
Measure: Mean (Standard Deviation); unit: Change in RV/LV Diameter Ratio
Arm/Group | Single Arm
Number analyzed (Participants) | 113
Change in RV/LV Diameter Ratio | 0.43 (0.26)

2. Primary Outcome: Major Adverse Event Rate
Description: A composite of: device-related death, major bleeding, device-related SAEs (a composite of clinical deterioration, pulmonary vascular injury, cardiac injury)
Time Frame: within 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 119
Participants | 2

3. Secondary Outcome: Device-related Death Rate
Time Frame: within 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 119
Participants | 1

4. Secondary Outcome: Major Bleeding Rate
Time Frame: within 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 119
Participants | 2

5. Secondary Outcome: Clinical Deterioration Rate
Time Frame: within 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 119
Participants | 2

6. Secondary Outcome: Pulmonary Vascular Injury Rate
Time Frame: within 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 119
Participants | 2

7. Secondary Outcome: Cardiac Injury Rate
Time Frame: within 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 119
Participants | 0

8. Secondary Outcome: Any-cause Mortality
Time Frame: within 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 119
Participants | 3

9. Secondary Outcome: Device-related SAE Rate
Time Frame: within 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 119
Participants | 2

10. Secondary Outcome: Symptomatic PE Recurrence Rate
Time Frame: within 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 119
Participants | 0

ADVERSE EVENTS:
Time Frame: Within 30 days post-procedure
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 3/119
Serious Adverse Events (participants affected / at risk) | 13/119
Other Adverse Events (participants affected / at risk) | 56/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=119)
Cardio-respiratory Arrest (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Ventricular Tachycardia (Cardiac disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Vascular Access Site Haemorrhage (Injury, poisoning and procedural complications) | 1
Ovarian Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 1
Stroke in Evolution (Nervous system disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=119)
Anaemia (Blood and lymphatic system disorders) | 5
Arrhythmia (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 2
Atrial Flutter (Cardiac disorders) | 1
Extrasystoles (Cardiac disorders) | 1
Supraventricular Tachycardia (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Abnormal Faeces (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Crohn's Disease (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest Pain (General disorders) | 4
Fatigue (General disorders) | 2
Hernia (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Vessel Puncture Site Pain (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Fungal Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Alcohol Poisoning (Injury, poisoning and procedural complications) | 3
Contusion (Injury, poisoning and procedural complications) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Head Injury (Injury, poisoning and procedural complications) | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1
Vascular Access Site Hemorrhage (Injury, poisoning and procedural complications) | 2
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 1
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Unresponsive To Stimuli (Nervous system disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 3
Haematuria (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Infarction (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1
Sputum Discoloured (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT03218566/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT03218566/SAP_001.pdf